CLINICAL TRIAL: NCT05213663
Title: Investıgatıon Of The Awareness Of The Parents Of The Cerebral Palsy Children About The Disease, Physiotherapy And Rehabilitation
Brief Title: Investıgatıon Of The Awareness Of The Parents Of Cerebral Palsy Children
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSUFTR
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Cerebral Palsy; Parents; Awareness; Physical Disability; Parenting
Keywords: parents; Awareness; physiotherapy and rehabilitation; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/parents of the Cerebral Palsy children: parents of the children with cerebral palsy will be evaluated about the awereness of their children's disease, physical and social activities and physiotherapy and rehabilitation.
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — To examine the awareness of parents of Cerebral Palsy children about the disease, physiotherapy and rehabilitation.

SUMMARY:
Parents of Cerebral Palsy (CP) children participate in treatments, education services and general medical check-ups; They have many responsibilities such as the use of drugs, devices, educational materials. Therefore, involving parents of CP children in the rehabilitation process provides a stronger rehabilitation service for their children. In the studies, it was stated that the active participation of the parents in the physiotherapy and rehabilitation process increases the success rate of the treatment and the participation of the parents plays a key role for the success of the physiotherapy and rehabilitation.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) children have a different clinical picture that includes many diseases. Abnormal muscle tone, insufficiency of postural control, weakness of muscle strength, abnormal behavior patterns and sensory problems are common symptoms, especially motor impairment can be in these children. These symptoms cause orthopedic problems, deformity and developmental delay over time. Motor disorders may be accompanied by various problems such as cognitive disorders, sensory, speech, cognitive, communication and behavioral problems, epilepsy and secondary musculoskeletal system problems. Functional skills such as independent sitting, standing, walking, balance, coordination, and fine motor skills are affected in these children due to different damage of neuronal system. This negatively affects the independence of activity in the child's daily life. CP children's treatment; It is carried out by a multidisciplinary team of specialists, such as specialist physicians, physiotherapists, psychologists, social counselors, child neurologists, orthopedists, vision-hearing specialists, pediatricians, occupational therapists, special educators, orthotics technicians, and with the participation of parents. The most important element of the rehabilitation team is the parents. In the postnatal period, parents are the primary responsible persons for the care of the child. This responsibility increases even more in the child with CP. The motor activity loss and movement disorder that develops in a child increase the functional dependency of the child in his daily life and cause him to need more support. All family members are somehow involved in the health services provided to these children. Parents are constantly involved in the life of the CP children and become aware of their child's abilities and needs. Parents of children participate in treatments, education services and general medical check-ups; They have many responsibilities such as the use of drugs, devices, educational materials. Therefore, involving parents of children in the rehabilitation process provides a stronger rehabilitation service for their children. In the studies, it was stated that the active participation of the parents in the physiotherapy and rehabilitation process increases the success rate of the treatment and the participation of the parents plays a key role for the success of the physiotherapy and rehabilitation. Parental support contributes to health and well-being and influences the success of long-term rehabilitation. With the increasing importance of family-centered practices in recent years, parents have started to take an active part in rehabilitation studies by continuing the practices in the clinic at home and in the community. It is an increasingly important view that parents play an important role in the lives of CP children. The acceptance of family-oriented care and the emergence of new theories on motor development have affected the treatment approach to these children, and the practices have become more family and function-centered rather than child-centered. The aim of this study is to investigate the awareness of parents of CP children about the disease, sports and physiotherapy and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being the parents of children with cerebral palsy between the ages of 4-18
* Volunteering to participate in the study
* Having communication skills to answer the questions in the personal information form and the evaluation form.

Exclusion Criteria:

• Having any psychiatric diagnosis of parents

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The universe of the research will consist of the parents of children with cerebral palsy who can be reached, who receive active treatment in special education and rehabilitation centers.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
1/The awareness of parents of children with Cerebral Palsy (CP) about the disease, physiotherapy and rehabilitation | first day of assessment
  The awareness of parents of children with Cerebral Palsy (CP) about the disease, physiotherapy and rehabilitation will be assessed with a 50-question questionnaire prepared by the researcher.

SECONDARY OUTCOMES:
Demographic information of parents | first day of assessment
  Demographic information of parents will be recorded (age, gender, height, body weight).
Demographic information of the children | first day of assessment
  Demographic information of the children will be recorded (age, gender, height, body weight,physiotherapy and rehabilitation years, diagnosis duration of the disease).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice adıgüzel, PhD, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No